CLINICAL TRIAL: NCT00002570
Title: A Phase III Study of Immediate Versus Delayed Chemotherapy for Asymptomatic Advanced Colorectal Cancer
Brief Title: Immediate Compared With Delayed Chemotherapy in Advanced Colorectal Cancer Without Signs or Symptoms of Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO10; CAN-NCIC-CO10 (Other: PDQ); NCCTG-JCO10 (Other: NCCTG); NCI-V94-0463 (Other Grant/Funding Number: NCI); CDR0000063607 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluorouracil and folinic acid (Active Comparator)
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium
- Observation (No Intervention)

INTERVENTIONS:
Drug: fluorouracil — 425 mg/m2 IV by bolus injection daily for 5 consecutive days q 28 days
  Arms: Fluorouracil and folinic acid
Drug: leucovorin calcium — 20 mg/m2 IV - number of cycles is determined by patient and physician
  Arms: Fluorouracil and folinic acid

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which treatment regimen is more effective for colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of immediate with delayed fluorouracil plus leucovorin in treating patients with advanced colorectal cancer without signs or symptoms of disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival and quality of life in asymptomatic patients with advanced colorectal cancer randomized to immediate fluorouracil/leucovorin (5-FU/CF) vs. 5-FU/CF delayed until onset of symptoms.

OUTLINE: Randomized, unblinded study. Arm I: Single-Agent Chemotherapy with Drug Modulation. Fluorouracil, 5-FU, NSC-19893; with Leucovorin calcium, CF, NSC-3590. Arm II: Observation followed by Single-Agent Chemotherapy with Drug Modulation. Clinical observation until symptomatic; followed by 5-FU; with CF.

PROJECTED ACCRUAL: 144 patients will be entered over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed cancer of the colon or rectum that is locally advanced or metastatic Primary lesion was or is located in the large bowel as confirmed by endoscopy, radiology, or surgery Radiologic or clinical evidence of metastasis subsequent to resection does not require histologic or cytologic confirmation unless: Interval between primary surgery and development of metastasis is greater than 5 years OR Primary cancer was Dukes' A or B1 Ineligible for potentially curative therapy, e.g.: Surgical resection of a limited hepatic or pulmonary metastasis Irradiation of locally recurrent colon or rectal cancer No or minimal symptoms related to the cancer, i.e.: No persistent pain requiring regular narcotic analgesia No persistent fever greater than 38 degrees C No symptomatic bowel obstruction No persistent nausea requiring medication No weight loss of greater than 5 kg over the previous 3 months unless clearly not associated with the cancer (e.g., associated with surgery or intercurrent illness) Symptomatic relapse/metastases rendered asymptomatic by secondary surgery or radiotherapy are eligible provided the patient remains asymptomatic for at least 6 weeks following such treatment No CNS metastases No significant ascites, pleural effusion, or pericardial effusion

PATIENT CHARACTERISTICS: Age: Adult under 80 (i.e., of legal age to sign own informed consent according to institutional policy) Performance status: Karnofsky 90-100% ECOG 0 Hematopoietic: Granulocytes at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal Renal: Creatinine less than 2.26 mg/dL Cardiovascular: No arrhythmia Other: No infection No other medical condition that is uncontrolled or could be aggravated by the protocol therapy No prior or concurrent second cancer except: Nonmelanomatous skin cancer In situ cervical cancer No pregnant women Adequate contraception required of fertile patients Blood/body fluid analyses to determine eligibility and quality-of-life questionnaire completed within 14 days prior to randomization; imaging studies of sites of disease completed within 28 days prior to randomization

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease or local recurrence Prior fluorouracil-based or other adjuvant therapy allowed At least 6 months required between completion of therapy and documentation of metastasis or recurrence Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Surgery: Prior surgery allowed

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 1994-07-15 (Actual); Primary Completion 2000-11 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Survival | 8 years

SECONDARY OUTCOMES:
Quality of life | 8 years
Toxicity | 8 years
Time to progression | 8 years
response rate | 8 years
response duration | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada; Henry C. Pitot, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hummer A, Carlo W, Sullivan D, et al.: Extensive hepatic resection does not correlate with toxicity following adjuvant chemotherapy. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-526, 2002.
- [Result] Ackland SP, Jones M, Tu D, Simes J, Yuen J, Sargeant AM, Dhillon H, Goldberg RM, Abdi E, Shepherd L, Moore MJ. A meta-analysis of two randomised trials of early chemotherapy in asymptomatic metastatic colorectal cancer. Br J Cancer. 2005 Nov 28;93(11):1236-43. doi: 10.1038/sj.bjc.6602841. PMID 16265352